CLINICAL TRIAL: NCT06804096
Title: Efficacy and Safety of Faropenem in Bangladeshi Adult Patients With Community-Acquired Bacterial Pneumonia (CABP): A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Faropenem in Bangladeshi Adult Patients With Community-Acquired Bacterial Pneumonia (CABP)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Md. Alimur Reza (Industry)
Responsible Party: Sponsor-Investigator, Dr. Md. Alimur Reza, Director, Beximco Pharmaceuticals Ltd.
Organization: Beximco Pharmaceuticals Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEX2410001
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Pneumonia, Community-Acquired; Bacterial Pneumonia
Keywords: CABP; Faropenem
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia, Bacterial | interventions — fropenem; Amoxicillin-Potassium Clavulanate Combination; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1: Tab. Faropenem 200mg three times daily with standard care.
  Interventions: Drug: Faropenem
- Arm 2 (Active Comparator): Arm 2: Tab. Co-Amoxiclav 625mg three times daily and Tab. Clarithromycin 500mg two times daily with standard care.
  Interventions: Drug: Co-amoxiclav; Drug: Clarithromycin 500 mg

INTERVENTIONS:
Drug: Faropenem — Tab. Faropenem 200mg three times daily
  Arms: Arm 1
Drug: Co-amoxiclav — Tab. Co-Amoxiclav 625mg three times daily
  Arms: Arm 2
Drug: Clarithromycin 500 mg — Tab. Clarithromycin 500mg two times daily
  Arms: Arm 2

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of faropenem in comparison to co-amoxiclav and clarithromycin in Bangladeshi adults diagnosed with community-acquired bacterial pneumonia (CABP). Eligible participants will be randomly assigned to one of two treatment arms. The first arm will receive faropenem at a dosage of 200 mg administered three times daily for a duration of seven days. The second arm will receive co-amoxiclav 625 mg, also three times daily, along with clarithromycin 500 mg, administered twice daily for seven days. All participants included in the study will undergo follow-up assessments over a period of four weeks. This research aims to provide valuable insights regarding the potential role of faropenem, thereby enhancing clinical outcomes and informing antibiotic stewardship in a region significantly burdened by CABP and characterized by limited treatment alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 to 65 years.
* Have an acute illness (less than or equal to 7 days duration) with any of the following signs and symptoms consistent with a lower respiratory tract infection (new or worsening):

  1. Fever (body temperature > 38.0 °C (100.4 °F) measured orally)
  2. Shortness of breath
  3. New onset or increased cough with or without sputum production.
  4. Chest pain.
* Have radiographically documented bacterial pneumonia:

  1. Infiltrates in a unilateral, lobar distribution
  2. Diffuse opacities or white condensed area
  3. The alveoli fill with white inflammatory fluid

Exclusion Criteria:

* Patients with severe pneumonia (Clinical & Radiological Assessment)
* Patients with suspicion of viral pneumonia (bilateral, patchy opacities, etc., in chest radiography.)
* Patients with suspicion of nosocomial pneumonia, aspiration pneumonia, etc.
* History of hypersensitivity, known or suspected contraindications, or intolerance to any of the study drugs.
* Intake of an antibiotic within the last 48 hours before study admission.
* History of hospitalization within the last 28 days.
* Patients in pregnancy and lactational state.
* Patients with Renal impairment (screening eGFR < 30mL/min).
* Significant hepatic impairment (Alanine aminotransferase > three times the upper limit of normal).
* Serious diseases that affect the immune system, such as Acquired Immunodeficiency Syndrome (AIDS), cancer, etc.
* Patients who are taking steroid medications, at least 20 mg daily dose of prednisolone (or equivalent doses of other glucocorticoids).
* Patients who are accepting chemotherapy or anti-cancer therapy or plan to receive such treatment during the trial or six months prior to enrollment.
* Had epilepsy, stroke, or other central nervous system disorders or uncontrolled psychiatric history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Cure Rate between two groups. | 10-14 days
  The clinical cure rate will be defined as significant improvement of clinical signs and symptoms at the end of treatment or follow-up, without new onset of symptoms, any complications, or the need for further antimicrobial therapy.
Percentage of patients withdrawn from the study due to adverse events between two groups. | 10-14 Days
  To compare the percentage of patients withdrawn from the study due to adverse events between two groups.

SECONDARY OUTCOMES:
Early Clinical Response (ECR) between two groups. | 3 - 4 days
  ECR will be defined as at least one improvement in the symptom mentioned below within 3 ± 1 days after the first dose of the study drug.
  1. Fever
  2. Decreased shortness of breath.
  3. Decreased chest pain.
  4. Decreased cough.
  5. Decreased sputum/mucous production.
  6. Sense of wellbeing.]
All-cause mortality between two groups | 10-14 days
  To compare the all-cause mortality rate between two groups
Number of patients who needed hospitalization in both groups | 28 days
Number of patients who needed Intensive Care Unit (ICU) support in both groups. | 28 Days
Frequency of Adverse Events & Serious Adverse Events between two groups. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Khan Abul Kalam Azad, Principal Investigator — Popular Medical College Hospital; Prof. Quazi Tarikul Islam, MBBS, FCPS, FACP (USA), FRCP,, Study Director — Popular Medical College Hospital
Locations (2):
- Bangladesh (2):
  - Popular Medical College & Hospital, Dhaka, Dhaka Division
  - Shaheed Suhrawardy Medical College & Hospital, Dhaka, Dhaka Division

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lode H, Magyar P, Muir JF, Loos U, Kleutgens K; International Gatifloxacin Study Group. Once-daily oral gatifloxacin vs three-times-daily co-amoxiclav in the treatment of patients with community-acquired pneumonia. Clin Microbiol Infect. 2004 Jun;10(6):512-20. doi: 10.1111/j.1469-0691.2004.00875.x. PMID 15191378
- [Background] Schurek KN, Wiebe R, Karlowsky JA, Rubinstein E, Hoban DJ, Zhanel GG. Faropenem: review of a new oral penem. Expert Rev Anti Infect Ther. 2007 Apr;5(2):185-98. doi: 10.1586/14787210.5.2.185. PMID 17402834
- [Background] Rudan I, Boschi-Pinto C, Biloglav Z, Mulholland K, Campbell H. Epidemiology and etiology of childhood pneumonia. Bull World Health Organ. 2008 May;86(5):408-16. doi: 10.2471/blt.07.048769. PMID 18545744
- [Background] Morens DM, Taubenberger JK, Fauci AS. Predominant role of bacterial pneumonia as a cause of death in pandemic influenza: implications for pandemic influenza preparedness. J Infect Dis. 2008 Oct 1;198(7):962-70. doi: 10.1086/591708. PMID 18710327
- [Background] Bartlett JG. Diagnostic tests for agents of community-acquired pneumonia. Clin Infect Dis. 2011 May;52 Suppl 4:S296-304. doi: 10.1093/cid/cir045. PMID 21460288
- [Background] Torres A, Peetermans WE, Viegi G, Blasi F. Risk factors for community-acquired pneumonia in adults in Europe: a literature review. Thorax. 2013 Nov;68(11):1057-65. doi: 10.1136/thoraxjnl-2013-204282. PMID 24130229
- [Background] Peto L, Nadjm B, Horby P, Ngan TT, van Doorn R, Van Kinh N, Wertheim HF. The bacterial aetiology of adult community-acquired pneumonia in Asia: a systematic review. Trans R Soc Trop Med Hyg. 2014 Jun;108(6):326-37. doi: 10.1093/trstmh/tru058. Epub 2014 Apr 29. PMID 24781376
- [Background] File TM Jr, Marrie TJ. Burden of community-acquired pneumonia in North American adults. Postgrad Med. 2010 Mar;122(2):130-41. doi: 10.3810/pgm.2010.03.2130. PMID 20203464
- [Background] Jain S, Self WH, Wunderink RG, Fakhran S, Balk R, Bramley AM, Reed C, Grijalva CG, Anderson EJ, Courtney DM, Chappell JD, Qi C, Hart EM, Carroll F, Trabue C, Donnelly HK, Williams DJ, Zhu Y, Arnold SR, Ampofo K, Waterer GW, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, McCullers JA, Pavia AT, Edwards KM, Finelli L; CDC EPIC Study Team. Community-Acquired Pneumonia Requiring Hospitalization among U.S. Adults. N Engl J Med. 2015 Jul 30;373(5):415-27. doi: 10.1056/NEJMoa1500245. Epub 2015 Jul 14. PMID 26172429